CLINICAL TRIAL: NCT04385355
Title: Influence of the Design of the Transmucosal Abutment on the Marginal Periimplant Bone Loss. Randomized Clinical Trial
Brief Title: Influence of the Design of the Transmucosal Abutment on the Periimplant Bone Level
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Santiago de Compostela (Other)
Collaborators: Mozo Grau Ticare Implants (Unknown)
Responsible Party: Principal Investigator, Juan Blanco Carrión, Professor, University of Santiago de Compostela
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ECRMGTCP2020
Record Dates: First submitted 2020-05-06; First posted 2020-05-12 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Peri-implant Marginal Bone Loss; Peri-implant Bone Level; Transmucosal Abutment Design; Peri-implant Bone Loss
Keywords: periimplant bone loss; abutment design; transmucosal abutment

STUDY DESIGN:
Intervention Model Description: For each participant on the test group will be another participant on the control group
Who Masked: Participant, Outcomes Assessor
Masking Description: None of the participants or the outcomes assessor will know the device (transmucosal abutment) received. The care provider will connect the transmucosal abutment while the surgery, after opening the randomization envelope; and the investigator will identify the participant's group while analysing the radiographs.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Other): Control group will receive an intermediate transmucosal abutment with conventional diameter and 3mm height, once the implants are placed.
  Interventions: Device: Conventional transmucosal abutment design
- Test Group (Experimental): Test group will receive an intermediate transmucosal abutment with a TCP design, narrower than the conventional one, of 3mm height, once the implants are placed
  Interventions: Device: Narrow transmucosal abutment design

INTERVENTIONS:
Device: Conventional transmucosal abutment design — The macroscopic design of the intermediate transmucosal abutment will be evaluated on terms of the marginal peri-implant bone levels using two identical devices, if only being the test device narrower than the control one
  Arms: Control Group
Device: Narrow transmucosal abutment design — The macroscopic design of the intermediate transmucosal abutment will be evaluated on terms of the marginal peri-implant bone levels using two identical devices, if only being the test device narrower than the control one
  Arms: Test Group

SUMMARY:
The objective of this study is to evaluate the radiographic changes on the marginal peri-implant bone level on bone level implants with a narrower transmucosal abutment, in comparison to the conventional abutment, both of 3mm height

DETAILED DESCRIPTION:
Patients will receive from one to eight bone-level implants according to their rehabilitation necessity and transmucosal abutments will be connected the day of the surgery. The control group will receive conventional transmucosal abutments while the test group will receive TCP abutments, with a narrower design.

Results will be evaluated initially 6 and 12 months after the connection of the definitive prostheses, and finally 3 years later.

ELIGIBILITY:
Inclusion Criteria:

* Absence of systemic and periodontal pathology, over 18 years of age, with a plaque index below 25%.
* Absence of at least one tooth, with natural adjacent teeth, allowing a prosthetic rehabilitation with an osseointegrated implant and a prosthetic unit.
* Adequate bone quality available, allowing placement of MOZO GRAU® implants InHex STD QUATTRO with diameters of 3.75 mm or 4.25 mm and lengths of 8, 10 and 11.5 mm.
* Natural teeth or implants with fixed restoration as antagonists.

Exclusion Criteria:

* Systemic factors:

  * Continuous administration of systemic medication that can interfere with the bone metabolism or medical conditions requiring prolonged use of steroids and / or medications that can interfere with bone metabolism.
  * History of leukocyte dysfunction and deficiency, immunodeficiency syndromes, kidney failure or bone metabolic disorders, such as osteoporosis.
  * Physical disability that may interfere with proper oral hygiene.
  * Use of any investigational medication or device within the previous 30 days to implant surgery in the study.
  * Alcoholism or drug addiction
  * Smoker of more than 10 cigarettes per day.
  * Conditions or circumstances that could prevent compliance with participation in study or interfere with the analysis of results, such as a history of breach or unreliability.

Local factors:

* History of local radiotherapy.
* Bruxism.
* Diseases that affect the oral mucosa, such as oral lichen planus.
* Untreated periodontitis.
* Persistent intraoral infection.
* Post-extraction alveoli not cured (less than 6 weeks after extraction).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Radiographic marginal periimplant bone level changes | from baseline (connection of the definitive abutment) to 6 and 12 months after the definitive prostheses will be connected, and finally 3 years later
  Measured as the distance from the bone crest to the first implant-to-bone contact. This will be assessed on parallelized periapical radiographies

SECONDARY OUTCOMES:
Probing pocket depth | 6 and 12 months after the definitive prostheses will be connected, and finally 3 years later
  measured with a CP12 probe as the distance from the soft tissue margin to the bottom of the peri-implant pocket
Papilla refill | 6 and 12 months after the definitive prostheses will be connected, and finally 3 years later
  Evaluated according to the Jemt 1997 index
Bleeding on probing | 6 and 12 months after the definitive prostheses will be connected, and finally 3 years later
  Evaluated according to the Mombelli 1987 index, presence of bleeding after probing
Plaque index | 6 and 12 months after the definitive prostheses will be connected, and finally 3 years later
  Evaluated according to the Mombelli 1987 index, presence of plaque
Patient Reported Outcomes Measurements | 6 and 12 months after the definitive prostheses will be connected, and finally 3 years later
  Using a visual analoge scale from 1 to 10 to evaluate patient's satisfaction parameters related to the aesthetics, masticatory ability, confort, general satisfaction and phonetics
Adverse effects frequency | 6 and 12 months after the definitive prostheses will be connected, and finally 3 years later
  Presence of adverse effects during the follow-up, such as fracture of the implant or the prosthetic unit or presence of periimplantitis or mucositis

CONTACTS AND LOCATIONS:
Locations (1):
- University of Santiago de Compostela, Santiago de Compostela, La Coruña, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alves CC, Munoz F, Cantalapiedra A, Ramos I, Neves M, Blanco J. Marginal bone and soft tissue behavior following platform switching abutment connection/disconnection--a dog model study. Clin Oral Implants Res. 2015 Sep;26(9):983-91. doi: 10.1111/clr.12385. Epub 2014 Apr 16. PMID 24735458
- [Background] Berglundh T, Lindhe J. Dimension of the periimplant mucosa. Biological width revisited. J Clin Periodontol. 1996 Oct;23(10):971-3. doi: 10.1111/j.1600-051x.1996.tb00520.x. PMID 8915028
- [Background] Blanco J, Pico A, Caneiro L, Novoa L, Batalla P, Martin-Lancharro P. Effect of abutment height on interproximal implant bone level in the early healing: A randomized clinical trial. Clin Oral Implants Res. 2018 Jan;29(1):108-117. doi: 10.1111/clr.13108. Epub 2017 Dec 8. PMID 29222809
- [Background] Ericsson I, Persson LG, Berglundh T, Marinello CP, Lindhe J, Klinge B. Different types of inflammatory reactions in peri-implant soft tissues. J Clin Periodontol. 1995 Mar;22(3):255-61. doi: 10.1111/j.1600-051x.1995.tb00143.x. PMID 7790533
- [Background] Koutouzis T, Adeinat B, Ali A. The influence of abutment macro-design on clinical and radiographic peri-implant tissue changes for guided, placed, and restored implants: A 1-year randomized controlled trial. Clin Oral Implants Res. 2019 Sep;30(9):882-891. doi: 10.1111/clr.13493. Epub 2019 Jun 24. PMID 31180160
- [Background] Novoa L, Batalla P, Caneiro L, Pico A, Linares A, Blanco J. Influence of Abutment Height on Maintenance of Peri-implant Crestal Bone at Bone-Level Implants: A 3-Year Follow-up Study. Int J Periodontics Restorative Dent. 2017 Sep/Oct;37(5):721-727. doi: 10.11607/prd.2762. PMID 28817138
- [Background] Souza AB, Alshihri A, Kammerer PW, Araujo MG, Gallucci GO. Histological and micro-CT analysis of peri-implant soft and hard tissue healing on implants with different healing abutments configurations. Clin Oral Implants Res. 2018 Oct;29(10):1007-1015. doi: 10.1111/clr.13367. Epub 2018 Sep 23. PMID 30246409